CLINICAL TRIAL: NCT06332443
Title: Randomized, Controlled Trial Comparing the Effectiveness of Sedation-Epidural Anesthesia to Spinal Anesthesia in Outpatient Hip or Knee Arthroplasty.
Acronym: RCT SEA vs SA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Mina Wahba Morcos (Unknown); Issam Tanoubi (Unknown); Pierre Drolet (Unknown); Ariane Clairoux (Unknown); Veronique Brulotte (Unknown); Marie-Eve Bélanger (Unknown); Philippe Richebé (Unknown); Karina Pellei (Unknown)
Responsible Party: Principal Investigator, Pascal André Vendittoli, Orthopedist, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER-CEMTL-2023-3086
Record Dates: First submitted 2024-03-14; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Knee Injuries and Disorders; Hip Injuries; Anesthesia
MeSH Terms: conditions — Knee Injuries; Disease; Hip Injuries | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: This study is a RCT with two parallel treatment groups: THA/TKA with single-shot SA group and THA/TKA with SED-EA group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The group assignment will be given to the intraoperative anesthesia team by writing, by a research team member who will not participate in postoperative assessments. The intraoperative anesthesia team will not be blinded to the group assignment, but surgeons, patients, and assessors will be blinded. For the SA group, a sham epidural catheter will be placed on the patient's back by the anesthesia team in order to keep the surgeons, patients and assessors blind to the randomization group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SA (Active Comparator): SA will be performed in the sitting or lateral position under sterile conditions. Spinal puncture will be performed at L2-L4 level using 50 mg of Clorotekal 1 or 2%. (intermediate-acting amide local anesthesia, commonly used) will be injected (32-34)
  Interventions: Procedure: Spinal anesthesia
- SED-EA (Active Comparator): EA will be performed in the sitting or lateral position under sterile conditions. Epidural puncture will be performed at the L2-L4 level and an epidural catheter will be inserted into the epidural space. 10 ml of 2% xylocaine without epinephrine will be injected through the catheter and the dose will be titrated (up to 20 mL) to achieve complete sensory block up to T12 dermatoma measured with a level to ice.
  Interventions: Procedure: Sedation epidural anesthesia

INTERVENTIONS:
Procedure: Spinal anesthesia — Spinal anesthesia will be performed in the sitting or lateral position under sterile conditions. Spinal puncture will be performed at L2-L4 level using 50 mg of Clorotekal 1 or 2%. (intermediate-acting amide local anesthesia, commonly used) will be injected.
  Arms: SA
Procedure: Sedation epidural anesthesia — Sedation-EA will be performed in the sitting or lateral position under sterile conditions. Epidural puncture will be performed at the L2-L4 level and an epidural catheter will be inserted into the epidural space. 10 ml of 2% xylocaine without epinephrine will be injected through the catheter and the dose will be titrated (up to 20 mL) to achieve complete sensory block up to T12 dermatoma measured with a level to ice.
  Arms: SED-EA

SUMMARY:
To our knowledge, no study has compared the difference between these two NA techniques. Early postoperative adverse events like uncontrolled pain, orthostatic hypotension, urinary retention, and prolonged motor block are linked to late patient mobilization, prolong hospitalization and failure to discharge in outpatient setting. The type of anesthesia used may have an important impact. Therefore, this study has the potential to improve the already established ERAS program and improve patients care perioperative and postoperative. Showing that SED-EA and SA are equivalent will allow for a more efficient and reliable technique for THA/TKA ERAS program that can be further translated into other lower limb surgeries.

DETAILED DESCRIPTION:
Primary objective is to compare the overall complication rate within 72 hours after surgery, categorized according to the Clavien-Dindo classification (15), between both techniques following THA and TKA surgery.

Secondary objectives are to compare the following perioperative and postoperative events between both groups:

1. Perioperative

   1. Preoperative pain levels and opioid/analgesics consumption
   2. Time needed to perform the technique (from the first handling the needle to sterile drapes removal from the back of the patient)
   3. Time needed for the SA or SED-EA to achieve adequate sensory block (from LA injection to the absence of cold feeling at T8 allowing surgical incision
   4. Intraoperative blood loss
   5. Need for dose adjustment intraoperatively
   6. Hemodynamic instability defined by hypotension (-20% from basal values prior to entering the OR, at the time of the consent).
2. Post-operative

   1. Time to motor and sensory function return
   2. Time to mobilization
   3. Pain evaluated with Visual analog scale immediately after surgery and up to 72 hours after surgery
   4. Opioid consumption up to 48 hours
   5. Hospital LOS and incidence of failed discharge at planned time
   6. Complications related to the technique performed (Post-dural puncture headache, local infection, hematoma etc.)

HYPOTHESIS We hypothesize that the incidence of the overall complication rate within 3 days after surgery, categorized according to the Clavien-Dindo classification will be equivalent between both groups; SED-EA and SA.

ELIGIBILITY:
Inclusion Criteria:

* Patient has symptomatic hip or knee OA requiring primary joint replacement (not associated with unusual treatments such as bone graft, concomitant osteotomy, revision implant, etc.).
* Patient who is candidate for our ERAS program
* Patient understands the study condition
* Patient capable of giving informed consent.
* Someone to accompany the patient to the Pre-admission Clinic and hospital the day of the surgery and to be available in the first postoperative week during home recovery.

Exclusion Criteria:

* Patients with contraindication to NA (spinal anatomical abnormalities, coagulation disorders, infection at the puncture site)
* Allergy to LAs used in the study
* Unable to communicate with the investigators, unable to read the questionnaire, unable to keep track and notes of the medication taken at home
* Lack of home services offered by the local community service centre in the area.
* BMI > 40.
* Psychiatric disease limiting participation or interfering with the ability to provide consent or assessment
* Need for long-term urinary Foley catheter post-op.
* Allergies to sulfonamides or other medications specified in the protocol.
* Cognitive impairment or communication problem
* Pulmonary embolism or deep vein thrombosis in the past year.
* Need for long-term anticoagulation therapy.
* Current corticotherapy or systemic corticotherapy in the past year (unless confirmation of a cortrosyn test prior to surgery).
* Systemic disease involvement (diabetes, heart, kidney, blood, etc.) necessitating special perioperative care (intensive care, multiple transfusions, dialysis, etc.).
* Coagulation disorder increasing the risk of intraoperative and postoperative bleeding including thrombocytopenia (platelet count lower than 80), hemophilia, prolonged INR (1,4 and over) and any order coagulation disorder deemed a contra-indication to neuraxial anesthesia..
* Locomotor problem, other than the joint to be replaced, imposing functional limitations that prevent movement without technical or physical assistance.
* Neurological or balance disorder.
* Living space incompatible with home care.
* Clcr < 30 ml/min (Cockcroft-Gault formula).
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Day 3
  The number of overall adverse events will be categorized according to the Clavien-Dindo classification

SECONDARY OUTCOMES:
Time needed by the anesthesiologist to perform the technique | Day 0
  Defined as the time frame from the end of the disinfection process to the time the medication is injected in the SA group or the catheter is secure in the SED-EA group (unit: mins).
Time needed for the SA or SED-EA to achieve adequate sensory block | Day 0
  defined as the time frame from the end of the anesthesia technique to the time the patient can no longer feel cold at her lower extremity.
Intraoperative blood loss | Day 0
  measured from the contents of suction bottles and the increased weight of surgical swabs by the operative nurse.
intraoperative muscle tension | Day 0
  rating which is rated on 4-point scale that blinded surgeons will use. The scale is as follows: 0 = most relaxed; 1 = mildly tight; 2 = moderately tight; and 3 = very tight.
Extra Lidocaine needed | Day 0
  An extra 5 mL of lidocaine 2% will be administrated through the SED-EA catheter if muscle tension or analgesia is judged not optimal by the surgeon and/or anesthesiologist. Need for dose adjustment of the SED-EA intraoperatively will be recorded by the anesthetist.
Conversion to GA | Day 0
  If muscle tension and/or analgesia is still deemed suboptimal with extra lidocaine in SED-EA of after a SA, conversion to GA will be accomplished using propofol, remifentanil and a neuromuscular blocking agent. No IV opioids will be used. Anesthesia maintenance will be performed with TIVA. Rate of conversion to GA will be recorded by research personnel.
Total dose of the sedation | Day 0
  Propofol sedation will be adjusted to keep a BIS index value in between 60 and 80.
Hemodynamic stability measured | Day 0
  All hemodynamic parameters will be recorded by a computer hooked onto the anesthesia monitors. A mean arterial pressure (MAP) of 70 mmHg or higher will be kept with phenylephrine in 100 mcg increments (if heart rate (HR) of 50/minute and over) or ephedrine in 5 mg increments (if HR under 50). Total doses of vasopressors used will be recorded.
Time to return of motor and sensory function | Day 1
  time to return of motor function is defined as the time when muscle strength in all three muscle groups tested is 5 of 5 on a 0 to 5 scale. The sensory dermatome level will be assessed using ice at the time of motor function return. Both assessments will begin 30 minutes after PACU arrival and continue every 30 minutes until motor function returns.
Post-operative nausea | Day 1
  Post-operative nausea and vomiting (PONV), dizziness and confusion will be recorded by the PACU nurse using Aldrete scores.
PONV and anti-emetics | Day 1
  PONV and anti-emetics in day care unit will be recorded.
Urinary retention | Day 1
  Urinary retention, defined by the inability to urinate for 8 hours after surgery or the need for a placement of a straight catheter or foley, consistent with a previous study.
Opioid consumption | Day 2
  Opioid consumption will be collected by the research team.
Length of stay | Day 2
  Defined as the time frame from the end of the THA/TKA surgery to the time of the discharge order.
Failed discharded | Day 2
  Defined as patient who is unable to be discharged within 24 hours after the end of surgery.
Complications related to the technique performed. | Day 3
  Complications related to the technique performed.
Adverse event | Day 3
  Adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Mina Morcos, Dr, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Hopital Maisonneuve Rosemont, Montreal, Quebec, Canada